CLINICAL TRIAL: NCT02862782
Title: Combination of Gonadotropin-releasing Hormone Agonist and Human Chorionic Gonadotropin Triggered by Normal Responder in GnRH-antagonist Cycles
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0317-16-TLV
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: In-vitro Fertilization
MeSH Terms: interventions — Chorionic Gonadotropin; Gonadotropin-Releasing Hormone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hCG (Experimental): Injection of hCG - Human Chorionic Gonadotropin (Ovitrelle 250 mcg mcg - Merck Serono)
  Interventions: Drug: hCG (Ovitrelle 250 mcg mcg - Merck Serono)
- hCG + GnRH agonist (Experimental): Injection of hCG - Human Chorionic Gonadotropin (Ovitrelle 250 mcg mcg - Merck Serono) and GnRH agonist - Gonadotropin - releasing hormone (Decapeptyl 0.2mg - Ferring Gmgh)
  Interventions: Drug: hCG (Ovitrelle 250 mcg mcg - Merck Serono) + GnRH agonist (Decapeptyl 0.2mg - Ferring Gmgh)

INTERVENTIONS:
Drug: hCG (Ovitrelle 250 mcg mcg - Merck Serono)
  Arms: hCG
Drug: hCG (Ovitrelle 250 mcg mcg - Merck Serono) + GnRH agonist (Decapeptyl 0.2mg - Ferring Gmgh)
  Arms: hCG + GnRH agonist

SUMMARY:
Background

The trigger for the final maturation of the ovum by providing integration of Human Chorionic Gonadotropin (hCG) and Gonadotropin - releasing hormone (GnRH) agonist was first introduced long ago, but clinically not accepted until the advent of GnRH antagonist protocol in IVF treatment.

In a recently published work which compared two types of ovulation induction (standard dose of hcg and in combination of GnRH agonist) in women with normal ovarian response, there was a statistically significant increase in the rates of implantation, clinical pregnancies and live births rates by providing integration of hCG and GnRH agonist.

To conclude, providing GnRH agonist in combination of hCF in standard dose is today an accepted treatment for final maturation of the ovums.

OBJECTIVE

The investigators objective is to investigate whether providing integrated treatment of Gonadotropin - releasing hormone (GnRH) Agonist and human Chorionic Gonadotropin (hCG) to final maturation of the ovum can improve the quality of the embryos, clinical pregnancies and live births rates in women treated with GnRH Antagonist protocol.

The main objective is to compare between two existing treatments.

DETAILED DESCRIPTION:
Background

The trigger for the final maturation of the ovum by providing integration of Human Chorionic Gonadotropin (hCG) and Gonadotropin - releasing hormone (GnRH) agonist was first introduced long ago, but clinically not accepted until the advent of GnRH antagonist protocol in IVF treatment.

In order to prevent Ovarian Hyperstimulation Syndrome in the treatment cycles with GnRH antagonist protocol, it is possible to make the final maturation of the ovums by providing GnRH agonist.

In a recently published work which compared two types of ovulation induction (standard dose of hcg and in combination of GnRH agonist) in women with normal ovarian response, there was a statistically significant increase in the rates of implantation, clinical pregnancies and live births rates by providing integration of hCG and GnRH agonist.

To conclude, providing GnRH agonist in combination of hCF in standard dose is today an accepted treatment for final maturation of the ovums.

OBJECTIVE

The investigators objective is to investigate whether providing integrated treatment of Gonadotropin - releasing hormone (GnRH) Agonist and human Chorionic Gonadotropin (hCG) to final maturation of the ovum can improve the quality of the embryos, clinical pregnancies and live births rates in women treated with GnRH Antagonist protocol.

The main objective is to compare between two existing treatments.

PATIENTS & METHODS

Women treated through IVF by protocol Gnarl - Antagonist

ELIGIBILITY:
Inclusion Criteria:

* Women who are going through IVF by protocol GnRH - Antagonist

Exclusion Criteria:

* Women with Ovarian Hyperstimulation Syndrome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancies rate | 1 month
  Number of pregnancies per treatment Injection of hCG - Human Chorionic Gonadotropin (Ovitrelle 250 mcg mcg - Merck Serono) and GnRH agonist - Gonadotropin - releasing hormone (Decapeptyl 0.2mg - Ferring Gmgh) in comperesment to Human Chorionic Gonadotropin (Ovitrelle 250 mcg mcg - Merck Serono)

CONTACTS AND LOCATIONS:
Overall Officials: Beni Almog, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No